CLINICAL TRIAL: NCT03142737
Title: Are the "ounce-equivalents" in the Protein Foods Groups Really Equivalent?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 205366
Record Dates: First submitted 2017-05-02; First posted 2017-05-05 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2019-06

CONDITIONS: Protein Metabolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Red kidney bean intake (Experimental): Subjects will consume 1/2 cup of cooked red kidney bean following diet normalization for 3 days.
  Interventions: Other: Red kidney bean intake
- Eggs intake (Experimental): Subjects will consume 2 cooked large eggs following diet normalization for 3 days.
  Interventions: Other: Eggs intake
- Peanut butter intake (Experimental): Subjects will consume 2 tablespoons of peanut butter following diet normalization for 3 days.
  Interventions: Other: Peanut butter intake
- Ground beef intake (Experimental): Subjects will consume 2 ounces of 90% lean ground beef following diet normalization for 3 days.
  Interventions: Other: Ground beef intake
- Intact beef intake (Experimental): Subjects will consume 2 ounces of intact beef following diet normalization for 3 days.
  Interventions: Other: Intact beef intake

INTERVENTIONS:
Other: Red kidney bean intake — Each participant will consume 1/2 cup of cooked red kidney bean
  Arms: Red kidney bean intake
Other: Eggs intake — Each participant will consume 2 cooked large eggs.
  Arms: Eggs intake
Other: Peanut butter intake — Each participant will consume 2 tablespoons of peanut butter.
  Arms: Peanut butter intake
Other: Ground beef intake — Each participant will consume 2 ounces of 90% lean ground beef.
  Arms: Ground beef intake
Other: Intact beef intake — Each participant will consume 2 ounces of intact beef.
  Arms: Intact beef intake

SUMMARY:
The investigators will determine effects of different sources of protein on whole-body net protein synthesis and muscle protein synthesis in young healthy participants.

DETAILED DESCRIPTION:
Over the past 35 years the United States Department of Agriculture (USDA) Dietary Guidelines for Americans (DGAs) has sought to translate recommendations on nutrient requirements (i.e., Recommended Dietary Allowances (RDAs) from the Food and Nutrition Board of the Institute of Medicine (IOM) into practical nutritional advice for the American public. Over the same time interval in which the Dietary Guidelines have existed the occurrence of nutrition-related health problems in the United States has escalated dramatically, showing that the population of obesity in U.S. has reached to a total of 35.8%. In addition, the lack of appropriate focus on protein nutrition is a major shortcoming of the DGAs. Not only is the amount of protein not a major focus, but also absolutely no mention is made of protein quality. Protein quality refers to the amount, profile, and true ileal digestibility of the essential amino acids (EAAs) in the protein. However, the concept of protein quality is not new, as the Protein Digestible Corrected Amino Acid Score was published by the Food and Agriculture Organization of the World Health Organization in 1993. Although animal protein (and beef specifically) has much higher the Digestible Indispensable Amino Acid Score (DIAAS) than plant proteins, often by as much as two fold, DIAAS has not taken account of the importance of the amount and profile of EAAs in individuals proteins. Moreover, the misrepresentation of the equivalencies of various food sources of protein in MyPlate raises the question of the process by which this occurred, and how can the process be influenced to more accurately reflect that high quality of animal proteins, including beef? Therefore, we propose to make these measurements in response to intake of "equivalent "(according to MyPlate) amounts of beef, kidney beans, eggs and peanut butter. Demonstration that the functional responses to these varied sources of protein coincide with the predictions from the USDA nutrient data base and calculation of the DIAAS will provide needed support to redefine "ounce equivalents" of protein food sources according to those data bases for all animal and plant sources of protein.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 20-40 years
* BMI from 20 to 29.9 kg/m2

Exclusion Criteria:

* Current diagnosis of diabetes
* History of malignancy in the 6 months prior to enrollment
* History of gastrointestinal bypass surgery
* History of a chronic inflammatory condition or other chronic diseases (Lupus, HIV/AIDS, etc)
* Female subjects who are currently pregnant
* Subjects who are unable to eat animal protein
* Subjects who are unable to stop eating protein or Amino Acid (AA) supplements during the participation
* Subjects who report regular resistance training (more than twice per week)
* Subjects who have concomitant use of corticosteroids (ingestion, injection or transdermal)
* Hemoglobin less than 9.5 g/dL at the screening visit
* Platelets less than 250,000 at the screening visit.
* Any other disease or condition that would place the subject at increased risk of harm if they were to participate, at the discretion of the study physician

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2018-03-06 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Net protein synthesis rate | Up to 8.5 hours
  Net protein synthesis rate is determined in the 4.5-hour basal fasted period and 4-hous post-meal period over the 8.5-hour experimental period

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wolfe, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No